CLINICAL TRIAL: NCT03647982
Title: Open-Label, Active Controlled, Single-Center, Phase 1 Study to Determine the Anhidrotic Area and Safety of MEDITOXIN in Healthy Male Volunteers
Brief Title: Anhidrotic Area and Safety of MEDITOXIN in Healthy Male Valunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT01-KR17PAH110
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Anhidrotic Area; Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- botulinum toxin 1U (Experimental)
  Interventions: Drug: Meditoxin; Drug: Botox
- botulinum toxin 3U(25U/1ml) (Experimental)
  Interventions: Drug: Meditoxin; Drug: Botox
- botulinum toxin 5U (Experimental)
  Interventions: Drug: Meditoxin; Drug: Botox
- botulinum toxin 10U (Experimental)
  Interventions: Drug: Meditoxin; Drug: Botox
- botulinum toxin 3U(50U/1ml) (Experimental)
  Interventions: Drug: Meditoxin; Drug: Botox
- botulinum toxin 3U(12.5U/1ml) (Experimental)
  Interventions: Drug: Meditoxin; Drug: Botox

INTERVENTIONS:
Drug: Meditoxin — injection of MEDITOXIN into the intradermal of each contralateral upper back in equal doses
Drug: Botox — injection of Botox into the intradermal of each contralateral upper back in equal doses

SUMMARY:
To determine the anhidrotic area and safety of MEDITOXIN

ELIGIBILITY:
Inclusion Criteria:

* Male adults aged between 20 and 45 years

Exclusion Criteria:

* Subjects not appropriate for participating in this study according to the investigator's opinion

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
anhidrotic area | week 4
  After the ninhydrin sweat test, measure the area of the unstained area

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University St. Paul Hospital, Seoul, Dongdaemun-gu, South Korea